CLINICAL TRIAL: NCT06377293
Title: Effects of Dialysis-specific Therapeutic Diet in Dialysis Patients
Brief Title: Effect of Dialysis-specific Therapeutic Diet on Biochemical Parameters in Dialysis Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Wan-Chuan Tsai, Principal Investigator, Assistant Professor, Far Eastern Memorial Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: FEMH-IRB-TSAI2024
Record Dates: First submitted 2024-04-15; First posted 2024-04-22 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: End-Stage Kidney Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: A randomized, active-controlled trial with cross-over design
Who Masked: Outcomes Assessor
Masking Description: Laboratory technicians who assess the study outcomes will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study diet (Experimental): 4-week therapeutic diet intervention as experimental group
  Interventions: Other: Dialysis-specific therapeutic diet
- Usual diet (No Intervention): 4-week usual diet as control group, no dietary intervention in this group, participants consumed their habitual diet

INTERVENTIONS:
Other: Dialysis-specific therapeutic diet — A healthy diet for dialysis patients
  Arms: Study diet

SUMMARY:
In patients with kidney failure, disturbances in bone turnover, mineral metabolism, vascular calcification, uremia, inflammation, immunity, metabolomics, nutrition, and gut microbial metabolites are frequent. Unhealthy diet causes altered mineral metabolism, elevated uremic toxin level, immune dysregulation, metabolic abnormalities, inflammation, protein-energy wasting and dysbiosis. The investigators hypothesize that therapeutic diet intervention reverses these uremic complications and thereby reduces cardiovascular risk in patients with kidney failure. In this study, the investigators crafted 4-week dialysis-specific therapeutic diet to illustrate the clinical implications of therapeutic diet for dialysis patients.

DETAILED DESCRIPTION:
In patients with kidney failure, disturbance in bone turnover and mineral metabolism, and nutritional deficiency is prevalent, leading to vascular calcification, uremia, inflammation, immune dysregulation, metabolic alteration, and gut microbial dysbiosis, and these abnormalities are associated with increased risk of fracture, extraskeletal or vascular calcification and cardiovascular mortality. It is well known that an unhealthy diet plays an important role in bone-mineral metabolism, uremia, inflammation, metabolomics, protein-energy wasting, and dysbiosis, and therefore nutritional therapy may help to manage these uremic complications to reduce cardiovascular risk in patients with kidney failure. Importantly, serum biomarkers regarding the above-mentioned abnormalities are acutely and closely related to food intake. To our knowledge, no study to date has examined the multifactorial effects of nutritional intervention on bone turnover, mineral metabolism, vascular calcification, uremia, inflammation, immunity, metabolomics, nutrition, and gut microbial metabolites in dialysis patients.

To examine the beneficial effects of nutritional intervention on clinical outcomes, the investigators crafted the dialysis-specific therapeutic diet which was characterized by adequate calorie and protein amounts, natural food ingredients with a low phosphorus-to-protein ratio, higher portions of plant-based food, and high fiber content. In the previous studies, the investigators found that the therapeutic diet rapidly reversed mineral abnormalities within the 1-week intervention period. Among these changes, reduction in serum phosphate level achieved in 2 days, modifications of intact parathyroid hormone (PTH) and calcium levels in 5 days, and reductions in intact and C-terminal fibroblast growth factor-23 (FGF23) levels in 7 days of therapeutic diet intervention. Although the therapeutic diet tended to change uremic toxin level, neither inflammatory nor nutritional markers changed which may be explained by short duration of intervention. It is of interest to know whether the therapeutic diet has a favorable effect on bone turnover, vascular calcification, and gut microbial dysbiosis. In this continuity planning, the investigators are therefore going to analyze the 4-week diet-induced changes in biomarkers regarding bone turnover, metabolites, vascular calcification, and gut microbial metabolites in addition to the previously assessed mineral metabolism, uremia, inflammation, immunity, and nutrition in dialysis patients.

This project aims to explore the multiple diverse effects of dialysis-specific healthy diet on the changes of bone turnover, mineral metabolism, vascular calcification, uremia, inflammation, immunity, metabolomics, nutrition, and gut microbial metabolites in dialysis patients. In contrast to the previous approaches, bone biomarkers for both of bone formation and bone resorption, vascular calcification biomarkers, and gut microbial metabolites will be comprehensively examined. Revealing a complex correlation between the nutritional factors and bone turnover, mineral metabolism, vascular calcification, uremia, inflammation, immunity, metabolomics, nutrition, and gut microbial dysbiosis, this project may shed light on understanding of diet-mediated bone-mineral and uremic homeostasis and uncover strategies of nutritional therapy. A better knowledge of diet-induced pathway on human body homeostasis may lead to new strategies for preventing fracture, vascular calcification or cardiovascular disease risk.

It is to conduct a randomized controlled trial with cross-over design at a dialysis unit of tertiary teaching hospital in Northern Taiwan. Subjects with aged older than 20 years, end-stage kidney disease (ESKD) undergoing maintenance dialysis for more than three months, having adequate dialysis and good dietary compliance will be included. Each participant will receive one study meal during the run-in period to give him or her the opportunity to assess whether he or she can successfully complete the study meals over the next 4 weeks, thus excluding participants who do not prefer the dietary intervention. Then, participants will be randomly assigned into two groups: group A and group B. Those in group A will receive study diet for 4 weeks, followed by 16-week washout period and then receive 4-week usual diet. The opposite order of diets will be prescribed in group B. The study meals are prepared in the hospital cafeteria. Dietary compositions of the study diets were analyzed before the start of the study. The study outcome measures are difference in change-from-baseline values of abnormal mineral metabolism, altered bone turnover, vascular calcification, uremic toxin production, immune dysregulation, metabolite alteration, nutrition, inflammation and gut microbial metabolites between the therapeutic diet and the usual diet.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with aged older than 20 years
* End-stage kidney disease (ESKD) undergoing maintenance dialysis for more than three months
* Must have adequate dialysis
* Good dietary compliance

Exclusion Criteria:

* Serum albumin level less than 2.5 g/dL
* Hospitalization within the past 4 weeks
* Prebiotics, probiotics, symbiotics or antibiotics use within the past 4 weeks
* History of psychiatric disorders
* Having mental retardation
* Those who dislike of the study meals
* Soft diet requirement
* Vegetarian

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Concentrations of intact fibroblast growth factor 23 (pg/mL) | 4 weeks
  Difference in change-from-baseline intact fibroblast growth factor 23 (pg/mL) between therapeutic diet and usual diet

SECONDARY OUTCOMES:
Concentrations of C-terminal fibroblast growth factor 23 (RU/mL) | 4 weeks
  Difference in change-from-baseline C-terminal fibroblast growth factor 23 (RU/mL) between therapeutic diet and usual diet
Concentrations of phosphate (mg/dL) | 4 weeks
  Difference in change-from-baseline phosphate (mg/dL) between therapeutic diet and usual diet
Concentrations of calcium (mg/dL) | 4 weeks
  Difference in change-from-baseline calcium (mg/dL) between therapeutic diet and usual diet
Concentrations of intact parathyroid hormone (pg/mL) | 4 weeks
  Difference in change-from-baseline intact parathyroid hormone (pg/mL) between therapeutic diet and usual diet
Concentrations of bone-specific alkaline phosphatase (μg/L) | 4 weeks
  Difference in change-from-baseline bone-specific alkaline phosphatase (μg/L) between therapeutic diet and usual diet
Concentrations of procollagen-type 1 N-terminal-propeptide (P1NP) (ng/mL) | 4 weeks
  Difference in change-from-baseline procollagen-type 1 N-terminal-propeptide (P1NP) (ng/mL) between therapeutic diet and usual diet
Concentrations of tartrate resistance acid phosphatase-5b (TRACP-5b) (mIU/ml) | 4 weeks
  Difference in change-from-baseline tartrate resistance acid phosphatase-5b (TRACP-5b) (mIU/ml) between therapeutic diet and usual diet
Concentrations of alkaline phosphatase (ALP) (IU/L) | 4 weeks
  Difference in change-from-baseline alkaline phosphatase (ALP) (IU/L) between therapeutic diet and usual diet
Concentrations of free indoxyl sulfate (mg/L) | 4 weeks
  Difference in change-from-baseline free indoxyl sulfate (mg/L) between therapeutic diet and usual diet
Concentrations of free p-cresol sulfate (mg/L) | 4 weeks
  Difference in change-from-baseline free p-cresol sulfate (mg/L) between therapeutic diet and usual diet
Concentrations of pre-albumin (g/dL) | 4 weeks
  Difference in change-from-baseline pre-albumin (g/dL) between therapeutic diet and usual diet
Concentrations of albumin (g/dL) | 4 weeks
  Difference in change-from-baseline albumin (g/dL) between therapeutic diet and usual diet
Concentrations of C-reactive protein (mg/dL) | 4 weeks
  Difference in change-from-baseline C-reactive protein (mg/dL) between therapeutic diet and usual diet
Concentrations of quinolinate | 4 weeks
  Difference in change-from-baseline quinolinate between therapeutic diet and usual diet
Concentrations of mesaconate | 4 weeks
  Difference in change-from-baseline mesaconate between therapeutic diet and usual diet
Absolute number (per μl blood) of CD4+ (cluster of differentiation 4) T cells | 4 weeks
  Difference in change-from-baseline absolute number (per μl blood) of CD4+ (cluster of differentiation 4) T cells between therapeutic diet and usual diet
Absolute number (per μl blood) of CD8+ (cluster of differentiation 8) T cells | 4 weeks
  Difference in change-from-baseline absolute number (per μl blood) of CD8+ (cluster of differentiation 8) T cells between therapeutic diet and usual diet
Absolute number (per μl blood) of monocytes | 4 weeks
  Difference in change-from-baseline absolute number (per μl blood) of monocytes between therapeutic diet and usual diet
Concentrations of fetuin-A (μg/ml) | 4 weeks
  Difference in change-from-baseline fetuin-A (μg/ml) between therapeutic diet and usual diet
Concentrations of trimethylamine-N-oxide (TMAO) (μM) | 4 weeks
  Difference in change-from-baseline trimethylamine-N-oxide (TMAO) (μM) between therapeutic diet and usual diet
Difference in change-from-baseline phosphate-binding equivalent dose (PBED) between therapeutic diet and usual diet | 4 weeks
  The phosphate-binder doses among the study participants will be compared by calculating the phosphate-binding equivalent dose (PBED) values as described by Daugirdas.

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Chuan Tsai, M.D., Ph.D., Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Banciao Dist., Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Individual-level deidentified participant data will be made available by the corresponding author of the paper upon request by email. The data will be available for 3 years after formal publication.
Supporting Information: Study Protocol
Time Frame: The data will become available after completing the study for 1 year and for 3 years after formal publication.
Access Criteria: Data will be made available by the corresponding author of the paper upon request by email.

REFERENCES:
- [Background] Tsai WC, Wu HY, Peng YS, Hsu SP, Chiu YL, Chen HY, Yang JY, Ko MJ, Pai MF, Tu YK, Hung KY, Chien KL. Effects of lower versus higher phosphate diets on fibroblast growth factor-23 levels in patients with chronic kidney disease: a systematic review and meta-analysis. Nephrol Dial Transplant. 2018 Nov 1;33(11):1977-1983. doi: 10.1093/ndt/gfy005. PMID 29420827
- [Background] Tsai WC, Peng YS, Wu HY, Hsu SP, Chiu YL, Liu LC, Tsai SM, Chien KL. Accuracy of a Nutrient Database in Estimating the Dietary Phosphorus-to-Protein Ratio and Using a Boiling Method in Low-Phosphate Hospital Diets. Sci Rep. 2018 Oct 15;8(1):15246. doi: 10.1038/s41598-018-33657-8. PMID 30323203
- [Background] Tsai WC, Wu HY, Peng YS, Hsu SP, Chiu YL, Yang JY, Chen HY, Pai MF, Lin WY, Hung KY, Chu FY, Tsai SM, Chien KL. Short-Term Effects of Very-Low-Phosphate and Low-Phosphate Diets on Fibroblast Growth Factor 23 in Hemodialysis Patients: A Randomized Crossover Trial. Clin J Am Soc Nephrol. 2019 Oct 7;14(10):1475-1483. doi: 10.2215/CJN.04250419. Epub 2019 Sep 13. PMID 31519550
- [Background] Tsai WC, Wu HY, Chiu YL, Yang JY, Pai MF, Wu YR, Lin WY, Hung KY, Chien KL, Hsu SP, Peng YS. Acute effects of dietary phosphorus intake on markers of mineral metabolism in hemodialysis patients: post hoc analysis of a randomized crossover trial. Ren Fail. 2021 Dec;43(1):141-148. doi: 10.1080/0886022X.2020.1870138. PMID 33427559
- [Background] Tsai WC, Hsu SP, Chiu YL, Wu HY, Luan CC, Yang JY, Pai MF, Lin CJ, Lin WY, Sun WH, Peng YS. Short-Term Effects of a Therapeutic Diet on Biochemical Parameters in Hemodialysis Patients: A Randomized Crossover Trial. J Ren Nutr. 2023 Nov;33(6):731-739. doi: 10.1053/j.jrn.2023.04.003. Epub 2023 Apr 27. PMID 37120127